CLINICAL TRIAL: NCT03610425
Title: A Standardized Bundle Protocol to Optimize Outcomes With Patients Undergoing Gynecological Surgery
Status: Completed | Type: Observational
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1088437
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-op evidence based bundle w/ Pre-op education: 25 patients undergoing hysterectomy from October 1, 2017 to December 31, 2017 will receive the post-operative evidence based bundle/standard pre-operative education.
- Standard pre-operative education alone: 25 patients undergoing hysterectomy from October 1, 2017 to December 31, 2017 will receive the standard pre-operative education alone.

SUMMARY:
Difference in outcome measures with the addition of post-operative evidence based bundle pre-operative education compared to standard pre-operative education given to patients prior to hysterectomy.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate whether there is a difference in outcome measures (length of stay, occurrence of readmission, and patient satisfaction) with the addition of a post-operative evidence-based bundle/standard pre-operative education compared to standard pre-operative education alone that is given to patients prior to a hysterectomy (open, vaginal, or laparoscopic).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted for all hysterectomies from October 1, 2017 through December 31, 2017, who speak English, and who are discharged home.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are admitted for all hysterectomies from October 1, 2017 through December 31, 2017, who speak English, and who are discharged home.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Length of Stay | 0 to 30 days
  Number of days spent in the hospital from the first post-operative day to the day of discharge
Occurrence of Re-Admission | 0 to 30 days
  Re-admission within 30 days will be measured through the EMR
Patient Satisfaction | 0 to 30 days
  Patient Satisfaction Survey that consists of 7 questions utilizing a likert scale from excellent to poor

CONTACTS AND LOCATIONS:
Locations (1):
- HonorHealth Scottsdale Thompson Peak, Scottsdale, Arizona, United States